CLINICAL TRIAL: NCT07016555
Title: Burning Mouth Syndrome: Symptoms and Management
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Alissa Nolden, Assistant Professor, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6052
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Burning Mouth Syndrome
Keywords: Symptom management; burning mouth syndrome; oral spray
MeSH Terms: conditions — Burning Mouth Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral spray (Experimental): Oral spray
  Interventions: Dietary Supplement: Oral cooling spray

INTERVENTIONS:
Dietary Supplement: Oral cooling spray — Use oral spray 3 times per day for 2 weeks

SUMMARY:
This research study aims to evaluate how an oral cooling spray, currently a commercial dietary supplement, impacts symptoms associated with burning mouth syndrome (BMS). This study will examine symptoms, frequency, and severity, along with other related side effects of BMS on food intake, enjoyment, and quality of life.

DETAILED DESCRIPTION:
Why are we doing this research study?

This research study aims to evaluate how an oral cooling spray, currently a commercial dietary supplement, impacts symptoms associated with burning mouth syndrome (BMS). This study will examine symptoms, frequency, and severity, along with other related side effects of BMS on food intake, enjoyment, and quality of life.

What are some of the important aspects of this research study that I should be aware of?

Timeframe: 2 weeks intervention

Use the oral cooling spray; "Dr.B's Elixir" as directed

Participants will report symptoms and other related impacts of BMS on a weekly online survey

Optional: complete a phone interview at the end of the 2-weeks intervention period (~30-60 minutes)

Optional: provide saliva samples (2 collections)

Compensation: No monetary compensation is provided

Direct benefit to research participants: Participants may experience changes in symptoms commonly experienced by BMS, but this is not guaranteed.

Who can participate in this research study?

We expect to enroll 30-50 individuals.

The eligibility criteria are:

At least 18 years old

Having been diagnosed with burning mouth syndrome or suffer from chronic oral burn without any identifiable causative lesion

No tongue or cheek piercings

No history of cancer

No recent or scheduled dental treatment

No history of gum disease

No aversions to mint or hop extracts

The exclusion criteria are:

Have recently undergone dental treatment in the last 3 months or have plans to undergo dental treatment (e.g., fillings, crowns, root canals, extractions, or other dental procedures) in the coming month.

Have started any new treatments for BMS in the last 3 months or have plans to start new treatments in the coming month.

What will I be asked to do, and how much time will it take?

The study will take place remotely in the comfort of your own home or residence. The study takes place over two weeks. Over the two weeks, you will use the oral spray 3 times per day with 5 sprays directly into your mouth on a single application and you can use up to 5 additional sprays as needed during each application. You will be completing an online questionnaire each week about symptoms related to BMS. This questionnaire is anticipated to take 5-10 minutes to complete. At the end of the 2nd week, participants have the option of participating in a phone interview which is anticipated to take approximately 30-60 minutes.

In total this is roughly an hour and a half if you participate in the entire study including the optional phone interview.

Optional: Phone interview

Participants have the option of participating in a phone interview - approximately 30-60 minutes at the end of the 2-weeks intervention period.

Optional: Salivary samples

Participants have the option to provide two salivary samples. The purpose of collecting saliva samples is to determine if the oral spray impacts the saliva composition compared to before its use. One sample will be collected before the oral cooling spray and one at the end of the two weeks. Then we will be doing shotgun metagenomics to analyze the total DNA content of the microbial community in the saliva samples. With this information, we can explore the oral microbiome which may be related to symptoms, taste, and flavor systems. For example, BMS has been associated with prevalent levels of "streptococcus", and it is expected that this oral spray may impact the levels of oral streptococcus.

Participants indicating consent to provide saliva samples will have saliva kits mailed along with the oral spray. After the end of the study, participants will drop the package in the mail. Return packaging and postage will be included. Participants will mail back the saliva kits with the pre-paid postage.

ELIGIBILITY:
Inclusion Criteria:

* Have buring mouth syndrome or experience oral burn
* Live in the United States
* At least 18 years old
* Having been diagnosed or suspected diagnosis of burning mouth syndrome or suffer from chronic oral burn without any identifiable causative lesion
* No tongue or cheek piercings
* No history of cancer
* No recent or scheduled dental treatment
* No history of gum disease
* No aversions to mint or hop extracts

Exclusion Criteria:

* Have recently undergone dental treatment in the last three months or have plans to undergo dental treatment (e.g., fillings, crowns, root canals, extractions, or other dental procedures) in the coming month.
* Have started any new treatments for BMS in the last 3 months or have plans to start new treatments in the coming month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Improved symptoms | 2 weeks
  Frequency, severity, and duration of oral burn between regular treatment decreases after 2 weeks of using the oral spray

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No